CLINICAL TRIAL: NCT02213809
Title: Effect of Case Method Education to General Practitioners on Their Knowledge on COPD and on the Health of Their Patients With COPD
Brief Title: Case Method Education on COPD to General Practitioners
Acronym: PRIMAIR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Dalarna County Council, Sweden (Other)
Responsible Party: Principal Investigator, Anna Nager, Senior lecturer and general practitioner, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2013/232-31/5
Record Dates: First submitted 2014-08-08; First posted 2014-08-12 (Estimated); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Case method education in COPD (Experimental): Two hours of case method education in COPD are given two times within 3 months to the general practitioners at nine primary health care centers. The education covers examination, including interpretation av spirometry, and treatment of patients with COPD. The learning outcomes are predefined and are the same in both arms. The same person will teach at both times of education.
  Interventions: Behavioral: Case method education in COPD
- Traditional education in COPD (Active Comparator): Two hours of traditional education in COPD are given two times within 3 months to the general practitioners at nine primary health care centers.The education covers examination, including interpretation av spirometry, and treatment of patients with COPD. The learning outcomes are predefined and are the same in both arms. The same person will teach at both times of education.
  Interventions: Behavioral: Traditional education in COPD

INTERVENTIONS:
Behavioral: Case method education in COPD — In case method a rich narrative describing of a real-life situation (teaching case) is presented, in which the learning group must make a decision or solve a problem. The teaching case provide information, but neither analysis nor conclusions. The analytical work of explaining the relationships among events in the case, identifying options, evaluating choices and predicting the effects of actions is the work done by students during the discussion.
  Arms: Case method education in COPD
Behavioral: Traditional education in COPD — Traditional education in this study means that the teacher mainly speaks to the group. Although short cases may be used for illustration, the main focus is not that the group shall solve problems from a narrative case.
  Arms: Traditional education in COPD

SUMMARY:
Background:

COPD is an inflammatory and chronic obstructive lung disease, mainly caused by smoking. Most patients with COPD are discovered and treated in primary health care. Co-morbidity with heart disease, hypertension, diabetes, osteoporosis and underweight is common. It is important to diagnose COPD at an early stage, primarily to motivate smoking cessation, which is the most important factor for decelerating the progress of COPD. In addition, medication and rehabilitation to reduce symptoms of COPD can be given. Previous studies in Sweden have shown poor quality of primary health care provided to patients with COPD.

As general practitioners often deal with multiple medical problems and patients' motivation when diagnosing and treating COPD we hypothesize that case method education (see description under "intervention") in COPD has better effect than traditional education (see description under "intervention").This study aims to examine the effect of case method education on (1) learning in COPD among general practitioners and on (2) health in their patients with COPD.

Method:

Primary health care centers (PHCC) in Stockholm will be recruited. The PHCCs will be randomized to either case method education (n=9 PHCCs) or traditional education (n=9 PHCCs) in COPD for their general practitioners. The educations will be held during two times (two hours each) within a time range of three months, covering examination and treatment of patients with COPD. At least 10.000 patients should be listed at PHCCs included. Random sampling of 45 patients with COPD at stage 2-3 will be done from each PHCC. The patients will fill in a self-assessment questionnaire including CCQ, CAT and LINQ (see outcome measures) as well as questions about medication, exacerbations and other chronic diseases. The questionnaire will be sent to the patients 1-2 months before the education and 18 months after the education. Differences in assessments in the questionnaire before and after the education will be compared between the patients listed at the PHCCs that have received case method education vs. traditional education. In addition, general practitioners (approximately, n=180) at the PHCCs will fill in a questionnaire, immediately before and 12 months after the education, covering the learning outcomes in order to study differences in learning between the two intervention groups.

ELIGIBILITY:
Inclusion Criteria:

* Primary Health Care Centers (PHCC): >10.000 patients listed. >70% permanent employed general practitioners
* Patients: Diagnosis of COPD registered at the COPD. Grade of COPD 2-3 (GOLD) at the latest spirometry completed since 2008.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 822 (Actual)
Dates: Start 2014-10-16 (Actual); Primary Completion 2018-12-12 (Actual); Study Completion 2018-12-12 (Actual)

PRIMARY OUTCOMES:
Difference i patients' assessment of Clinical COPD Questionnaire (CCQ) before the intervention and 18 months later. | 1-2 months before the intervention and 18 months after the intervention
  The CCQ measures health status in patients with COPD and consists of 10 items with an overall score and 3 domains: Symptoms (4 items), Functional state (4 items) and Mental state (2 items). All scores range from 0 to 6; (0 = no impairment).
Difference in questionnaire about knowledge in COPD (questionnaire created by the research group)among the general practitioners that receive the education. | Immediately before the intervention and 12 months later.
  The questionnaire covers examination and treatment of COPD and includes multiple choice questions as well as questions about attitudes that will be answered in free text.

SECONDARY OUTCOMES:
Difference i patients' assessment of Lung Information Needs Questionnaire (LINQ) before the intervention and 18 months later. | 1-2 months before the intervention and 18 months after the intervention
  LINQ measures patients perceptions about COPD and what information about COPD patients think that they have percieved from health care personnel.
Difference in patients' assessment of COPD Assessment Test (CAT) before the intervention and 18 months later. | 1-2 months before the intervention and 18 months after the intervention
  The COPD Assessment Test (CAT) measures the impact of COPD on a person's life.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Nager, PhD, Principal Investigator — Karolinska Institutet; Hanna Sandelowsky, MD, Study Director — Karolinska Institutet
Locations (1):
- Department of Family Medicine, NVS, Karolinska Institutet, Huddinge, Sweden

REFERENCES:
- [Derived] Sandelowsky H, Krakau I, Modin S, Stallberg B, Nager A. Primary care patients with mild or stable chronic obstructive pulmonary disease need more support in disease management: a secondary analysis of a cluster randomized controlled trial. Scand J Prim Health Care. 2023 Dec;41(4):495-504. doi: 10.1080/02813432.2023.2280039. Epub 2023 Nov 29. PMID 37975839
- [Derived] Sandelowsky H, Krakau I, Modin S, Stallberg B, Johansson SE, Nager A. Effectiveness of traditional lectures and case methods in Swedish general practitioners' continuing medical education about COPD: a cluster randomised controlled trial. BMJ Open. 2018 Aug 10;8(8):e021982. doi: 10.1136/bmjopen-2018-021982. PMID 30099398
- [Derived] Sandelowsky H, Krakau I, Modin S, Stallberg B, Nager A. Case Method in COPD education for primary care physicians: study protocol for a cluster randomised controlled trial. Trials. 2017 Apr 27;18(1):197. doi: 10.1186/s13063-017-1889-4. PMID 28449709